CLINICAL TRIAL: NCT00222482
Title: A Double-Blind and Placebo Controlled Assessment of Depakote ER in Borderline Personality Disorder
Brief Title: Depakote ER in Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Abbott (Industry); Schulz, S. Charles, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0306M49703; M009946
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2007-08-09 (Estimated); Status verified 2007-08

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Depakote ER

SUMMARY:
This study examines the effect of Depakote ER versus placebo in a randomized trial of borderline personality disorder. Patients all participate in DBT therapy and those who are not responsive are assigned to either Depakote ER or placebo for up to 12 weeks. Borderline Personality Symtoms are measured and side-effects are assessed.

ELIGIBILITY:
Inclusion Criteria:Male or female patients with the diagnosis of borderline personality disorder between the ages of 21 adn 55 years old. Must be in good physical health -

Exclusion Criteria:Major psychiatric illness on Axis I - schizophrenia or bipolar disorder. May not have current MDD. May not be dependent on illicit substances or alcohol.

-

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15
Dates: Start 2003-03; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Symptom Checklist 90

SECONDARY OUTCOMES:
Barratt Impulsivity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sellamnn C Schulz, M.D., Principal Investigator — Department of Psychiatry, University of Minnesota Medical School

REFERENCES:
- [Background] Schulz SC, Camlin KL, Berry SA, Jesberger JA. Olanzapine safety and efficacy in patients with borderline personality disorder and comorbid dysthymia. Biol Psychiatry. 1999 Nov 15;46(10):1429-35. doi: 10.1016/s0006-3223(99)00128-6. PMID 10578457
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174